CLINICAL TRIAL: NCT00989612
Title: Immunogenicity and Safety Study of GSK Biologicals' Influenza Candidate Vaccine GSK2340274A
Brief Title: Study to Evaluate Immunogenicity and Safety of an Investigational Influenza Vaccine (H1N1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113519
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: influenza infection; GSK Biologicals' influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- GSK2340274A GROUP (Experimental): Healthy subjects, aged 20 to 64 years, male and female, received 2 doses of GSK2340274A vaccine, injected intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
  Interventions: Biological: Influenza investigational vaccine GSK2340274A

INTERVENTIONS:
Biological: Influenza investigational vaccine GSK2340274A — Two intramuscular injections on Day 0 and Day 21, respectively

SUMMARY:
This trial will assess the immunogenicity and safety elicited by the adjuvanted GSK Biologicals' influenza investigational vaccine GSK2340274A in healthy Japanese adults aged 20-64 years.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol amendment 1& 2, October 2009. The sections impacted are study design and outcome measures

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female adults 20 to 64 years of age at time of the first vaccination, inclusive.
* Good general health as assessed by medical history and physical examination
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Females of non-childbearing potential may be enrolled in the study.
* Female of childbearing potential may be enrolled in the study, if she:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* History of previous administration of a novel [H1N1]v vaccine.
* Previous participation in study NCT00742885.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence or evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5 °C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Diagnosed with cancer, or treatment for cancer within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within 6 months of study enrolment or planned administration during the study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of any vaccines within 30 days before vaccination or planned administration within the first vaccination up to blood sampling at Day 42 and within 30 days prior to blood sampling at Day 182, with the exception of seasonal influenza vaccine.
* Administration of any seasonal influenza vaccine within 14 days before vaccination on Day 0, or planned administration within the first vaccination up to blood sampling at Day 42 and within 14 days prior to blood sampling at Day 182.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine test result prior to the time of first vaccination.
* Lactating or nursing female.
* Excessive underweight (Body Mass Index [BMI] < 18.5) or excessive obesity (BMI >= 30).
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10-01; Primary Completion 2010-04-19 (Actual); Study Completion 2010-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ikematsu H, Nagai H, Kawashima M, Kawakami Y, Tenjinbaru K, Li P, Walravens K, Gillard P, Roman F. Characterization and long-term persistence of immune response following two doses of an AS03A-adjuvanted H1N1 influenza vaccine in healthy Japanese adults. Hum Vaccin Immunother. 2012 Feb;8(2):260-6. doi: 10.4161/hv.18469. Epub 2012 Feb 1. PMID 22426369
- [Derived] Ikematsu H, Nagai H, Kawashima M, Kawakami Y, Tenjinbaru K, Maeda A, Li P, Gillard P, Roman F. Immunogenicity and safety of a novel AS03(A)-adjuvanted H1N1 2009 pandemic influenza vaccine in adults in Japan. Hum Vaccin. 2010 Nov;6(11):888-93. doi: 10.4161/hv.6.11.12851. Epub 2010 Nov 1. PMID 20980795
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113519 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2340274A Group
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 0
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects, who received the 2 vaccine doses and for whom assay results for antibodies against vaccine antigen were available.
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Titers | 8.8 [7.3 to 10.5]

2. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Titers | 230.3 [177.7 to 298.4]

3. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (97.5% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Titers | 485.0 [420.3 to 559.7]

4. Primary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies A/California/7/2009 (H1N1)V-like Antigen
Description: A seropositive subject was defined as a subject whose serum antibody titer was greater than or equal to (≥) 1:10.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 43

5. Primary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seropositive subject was defined as a subject whose serum antibody titer was greater than or equal to (≥) 1:10.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 100

6. Primary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seropositive subject was defined as a subject whose serum antibody titer was greater than or equal to (≥) 1:10.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 100

7. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer smaller than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 94

8. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: as for outcome 7
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 100

9. Primary Outcome: Number of Seroprotected Subjects Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 6

10. Primary Outcome: Number of Seroprotected Subjects Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 95

11. Primary Outcome: Number of Seroprotected Subjects Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 100

12. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (97.5% Confidence Interval); unit: Fold change
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Fold change | 26.3 [20.6 to 33.5]

13. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: as for outcome 12
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (97.5% Confidence Interval); unit: Fold change
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Fold change | 55.4 [45.6 to 67.2]

14. Secondary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies A/California/7/2009 (H1N1)V-like Antigen
Description: A seropositive subject was defined as a subject whose serum antibody titer was greater than or equal to (≥) 1:10.
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340274A 20-40Y Group: Healthy subjects, aged 20 to 40 years (Y), male and female, received 2 doses of GSK2340274A vaccine, injected intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
- GSK2340274A 41-64Y Group: Healthy subjects, aged 41 to 64 years (Y), male and female, received 2 doses of GSK2340274A vaccine, injected intramuscularly in the deltoid region of the non-dominant arm at Day 0 and of the dominant arm at Day 21.
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Participants
  Day 0 | 22 | 21
  Day 21 | 50 | 50
  Day 42 | 50 | 50
  Day 182 | 50 | 50

15. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Titers
  Day 0 | 8.9 [7.1 to 11.1] | 8.9 [6.8 to 10.9]
  Day 21 | 258.3 [191.3 to 348.7] | 205.3 [145.4 to 290.0]
  Day 42 | 505.6 [427.9 to 597.6] | 465.3 [384.5 to 563.0]
  Day 182 | 182.6 [141.1 to 236.4] | 167.9 [124.5 to 226.5]

16. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: as for outcome 7
Time Frame: At Days 21, 42 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Participants
  Day 21 | 50 | 44
  Day 42 | 50 | 50
  Day 182 | 48 | 45

17. Secondary Outcome: Number of Seroprotected Subjects Against A/California/7/2009 (H1N1)V-like Antigen
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Participants
  Day 0 | 3 | 3
  Day 21 | 50 | 45
  Day 42 | 50 | 50
  Day 182 | 49 | 46

18. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Antigen
Description: as for outcome 12
Time Frame: At Days 21, 42 and 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Fold change
  Day 21 | 29.1 [21.8 to 38.9] | 23.8 [17.4 to 32.6]
  Day 42 | 57.0 [44.3 to 73.2] | 53.9 [42.6 to 68.1]
  Day 182 | 20.6 [16.0 to 26.5] | 19.4 [15.1 to 25.1]

19. Secondary Outcome: Titers for Serum Neutralizing Antibodies Against A/Neth/602/09 (H1N1)V-like Antigen
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Titers
  Day 0 | 8.7 [6.6 to 11.4] | 8.4 [6.6 to 10.7]
  Day 21 | 146.6 [90.1 to 238.6] | 127.8 [77.1 to 211.9]
  Day 42 | 336.6 [247.8 to 457.1] | 277.7 [194.3 to 397.0]
  Day 182 | 133.5 [97.3 to 183.1] | 98.0 [66.6 to 144.3]

20. Secondary Outcome: Number of Seropositive Subjects for Neutralizing Antibodies Against A/Neth/602/09 (H1N1)V-like Antigen
Description: A seropositive subject was defined as a subject whose serum antibody titer was greater than or equal to (≥) 1:8.
Time Frame: At Days 0, 21, 42 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Participants
  Day 0 | 24 | 27
  Day 21 | 47 | 49
  Day 42 | 50 | 50
  Day 182 | 50 | 49

21. Secondary Outcome: Number of Seroconverted Subjects for Neutralizing Antibodies Against A/Neth/602/09 (H1N1)V-like Antigen
Description: A seroconverted subject was defined as a vaccinated subject with a minimum 4-fold increase in post vaccination neutralizing titer.
Time Frame: At Days 21, 42 and 182
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A 20-40Y Group | GSK2340274A 41-64Y Group
Number analyzed (Participants) | 50 | 50
Participants
  Day 21 | 39 | 35
  Day 42 | 48 | 48
  Day 182 | 42 | 34

22. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During a 7-day (Days 0-6) follow-up after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants
  Pain, Any, Dose 1 | 98
  Pain, Grade 3, Dose 1 | 3
  Redness, Any, Dose 1 | 7
  Redness, Grade 3, Dose 1 | 1
  Swelling, Any, Dose 1 | 17
  Swelling, Grade 3, Dose 1 | 2
  Pain, Any, Dose 2 | 93
  Pain, Grade 3, Dose 2 | 2
  Redness, Any, Dose 2 | 8
  Redness, Grade 3, Dose 2 | 0
  Swelling, Any, Dose 2 | 17
  Swelling, Grade 3, Dose 2 | 1
  Pain, Any, Across doses | 99
  Pain, Grade 3, Across doses | 5
  Redness, Any, Across doses | 13
  Redness, Grade 3, Across doses | 1
  Swelling, Any, Across doses | 24
  Swelling, Grade 3, Across doses | 2

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During a 7-day (Days 0-6) follow-up after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants
  Fatigue, Any, Dose 1 | 46
  Fatigue, Grade 3, Dose 1 | 2
  Fatigue, Related, Dose 1 | 45
  Headache, Any, Dose 1 | 35
  Headache, Grade 3, Dose 1 | 1
  Headache, Related, Dose 1 | 34
  Joint pain at other location, Any, Dose 1 | 14
  Joint pain at other location, Grade 3, Dose 1 | 0
  Joint pain at other location, Related, Dose 1 | 14
  Muscle aches, Any, Dose 1 | 44
  Muscle aches, Grade 3, Dose 1 | 1
  Muscle aches, Related, Dose 1 | 44
  Shivering, Any, Dose 1 | 19
  Shivering, Grade 3, Dose 1 | 0
  Shivering, Related, Dose 1 | 19
  Sweating, Any, Dose 1 | 7
  Sweating, Grade 3, Dose 1 | 0
  Sweating, Related, Dose 1 | 7
  Temperature (Axillary), Any, Dose 1 | 2
  Temperature (Axillary), Grade 3, Dose 1 | 0
  Temperature (Axillary), Related, Dose 1 | 2
  Fatigue, Any, Dose 2 | 54
  Fatigue, Grade 3, Dose 2 | 3
  Fatigue, Related, Dose 2 | 54
  Headache, Any, Dose 2 | 39
  Headache, Grade 3, Dose 2 | 2
  Headache, Related, Dose 2 | 37
  Joint pain at other location, Any, Dose 2 | 30
  Joint pain at other location, Grade 3, Dose 2 | 1
  Joint pain at other location, Related, Dose 2 | 30
  Muscle aches, Any, Dose 2 | 51
  Muscle aches, Grade 3, Dose 2 | 0
  Muscle aches, Related, Dose 2 | 51
  Shivering, Any, Dose 2 | 29
  Shivering, Grade 3, Dose 2 | 4
  Shivering, Related, Dose 2 | 29
  Sweating, Any, Dose 2 | 9
  Sweating, Grade 3, Dose 2 | 0
  Sweating, Related, Dose 2 | 9
  Temperature (Axillary), Any, Dose 2 | 7
  Temperature (Axillary), Grade 3, Dose 2 | 1
  Temperature (Axillary), Related, Dose 2 | 6
  Fatigue, Any, Across doses | 69
  Fatigue, Grade 3, Across doses | 5
  Fatigue, Related, Across doses | 68
  Headache, Any, Across doses | 51
  Headache, Grade 3, Across doses | 3
  Headache, Related, Across doses | 49
  Joint pain at other location, Any, Across doses | 33
  Joint pain at other location, Grade 3, Across dose | 1
  Joint pain at other location, Related, Across dose | 33
  Muscle aches, Any, Across doses | 59
  Muscle aches, Grade 3, Across doses | 1
  Muscle aches, Related, Across doses | 59
  Shivering, Any, Across doses | 37
  Shivering, Grade 3, Across doses | 4
  Shivering, Related, Across doses | 37
  Sweating, Any, Across doses | 13
  Sweating, Grade 3, Across doses | 0
  Sweating, Related, Across doses | 13
  Temperature (Axillary), Any, Across doses | 7
  Temperature (Axillary), Grade 3, Across doses | 1
  Temperature (Axillary), Related, Across doses | 6

24. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During a 21-day (Days 0-20) follow-up period after the first vaccination and during a 63-day (Days 21-84) follow-up after the second vaccination
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants
  Subjects with any AE(s) | 46
  Subjects with grade 3 AE(s) | 1
  Subjects with related AE(s) | 18

25. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (Days 0-182)
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 2

26. Secondary Outcome: Number of Subjects With Any Adverse Events of Specific Interest (AESIs).
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (Days 0-182)
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Participants | 0

27. Secondary Outcome: Number of Days With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. The number of days with any solicited local symptom was assessed in subjects who have reported at least once the symptom.
Time Frame: During a 7-day (Days 0-6) follow-up after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Median (Full Range); unit: Days
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Days
  Pain, Dose 1: number analyzed (Participants) | 98
  Pain, Dose 1 | 4 [1 to 7]
  Redness, Dose 1: number analyzed (Participants) | 7
  Redness, Dose 1 | 3 [1 to 6]
  Swelling, Dose 1: number analyzed (Participants) | 17
  Swelling, Dose 1 | 3 [1 to 7]
  Pain, Dose 2: number analyzed (Participants) | 93
  Pain, Dose 2 | 3 [1 to 7]
  Redness, Dose 2: number analyzed (Participants) | 8
  Redness, Dose 2 | 3 [1 to 6]
  Swelling, Dose 2: number analyzed (Participants) | 17
  Swelling, Dose 2 | 3 [1 to 7]

28. Secondary Outcome: Number of Days With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. The number of days with any solicited general symptom was assessed in subjects who have reported at least once the symptom.
Time Frame: During a 7-day (Days 0-6) follow-up after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects.
Measure: Median (Full Range); unit: Days
Arm/Group | GSK2340274A Group
Number analyzed (Participants) | 100
Days
  Fatigue, Dose 1: number analyzed (Participants) | 46
  Fatigue, Dose 1 | 2 [1 to 6]
  Headache, Dose 1: number analyzed (Participants) | 35
  Headache, Dose 1 | 1 [1 to 6]
  Joint pain at other location, Dose 1: number analyzed (Participants) | 14
  Joint pain at other location, Dose 1 | 2 [1 to 5]
  Muscle aches, Dose 1: number analyzed (Participants) | 44
  Muscle aches, Dose 1 | 3 [1 to 6]
  Sweating, Dose 1: number analyzed (Participants) | 7
  Sweating, Dose 1 | 1 [1 to 6]
  Shivering, Dose 1: number analyzed (Participants) | 19
  Shivering, Dose 1 | 1 [1 to 3]
  Temperature, Dose 1: number analyzed (Participants) | 2
  Temperature, Dose 1 | 1 [1 to 1]
  Fatigue, Dose 2: number analyzed (Participants) | 54
  Fatigue, Dose 2 | 2 [1 to 7]
  Headache, Dose 2: number analyzed (Participants) | 39
  Headache, Dose 2 | 1 [1 to 7]
  Joint pain at other location, Dose 2: number analyzed (Participants) | 30
  Joint pain at other location, Dose 2 | 2 [1 to 6]
  Muscle aches, Dose 2: number analyzed (Participants) | 51
  Muscle aches, Dose 2 | 3 [1 to 7]
  Sweating, Dose 2: number analyzed (Participants) | 9
  Sweating, Dose 2 | 1 [1 to 4]
  Shivering, Dose 2: number analyzed (Participants) | 29
  Shivering, Dose 2 | 1 [1 to 3]
  Temperature, Dose 2: number analyzed (Participants) | 7
  Temperature, Dose 2 | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7-day post-vaccination period (Days 0-6), Unsolicited AEs during the 31-day post-vaccination (Days 0-30), SAEs during the entire study period (Day 0 - Day 182).
Arm/Group | GSK2340274A Group
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 2/100
Other Adverse Events (participants affected / at risk) | 100/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340274A Group (N=100)
Calculus ureteric (Renal and urinary disorders) | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1
Viral infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340274A Group (N=100)
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 (44)
Chills (General disorders) | 37 (48)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 13 (15)
Fatigue (General disorders) | 69 (100)
Headache (Nervous system disorders) | 53 (79)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 59 (95)
Nasopharyngitis (Infections and infestations) | 5 (9)
Pain (General disorders) | 99 (191)
Pyrexia (General disorders) | 10 (13)
Swelling (General disorders) | 24 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.